CLINICAL TRIAL: NCT01894672
Title: A Phase 2 Trial of the BRAF Inhibitor, LGX818, Utilizing a Pulsatile Schedule in Patients With Stage IV or Unresectable Stage III Melanoma Characterized by a BRAFV600 Mutation
Brief Title: BRAF Inhibitor, LGX818, Utilizing a Pulsatile Schedule in Patients With Stage IV or Unresectable Stage III Melanoma Characterized by a BRAFV600 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-053
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2019-12

CONDITIONS: Melanoma
Keywords: LGX818; BRAF Inhibitor; Stage IV melanoma; unresectable stage III melanoma; BRAFV600 mutation; 13-053
MeSH Terms: conditions — Melanoma | interventions — encorafenib

ARMS (1):
- LGX818 (Experimental): LGX818 capsules will be administered orally on a once -daily schedule (QD) dosing at a dose of 300 mg/day, 2 weeks on followed by a 2 week break. This schedule of 2 weeks on, followed by 2 weeks off, will continue for the duration of time the patients remains on the clinical trial. After the follow up visit patients will be contacted approximately every 12 weeks until they have received a subsequent therapy or until they have been off treatment for a year to monitor their survival.
  Interventions: Drug: LGX818

INTERVENTIONS:
Drug: LGX818

SUMMARY:
The purpose of this phase II study is to find out if an investigational drug called LGX818 can stop the melanoma from growing.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV, or unresectable stage III melanoma that harbors a BRAFV600 mutation
* Any prior therapy allowed except a BRAF or MEK inhibitor,.
* Patients must provide written informed consent prior to any screening procedures.
* Age 18 years or older.
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Patient is able to swallow and retain oral medication
* Measurable disease according to RECIST v1.1
* ECOG performance status ≤ 1

Exclusion Criteria:

* Brain metastasis or leptomeningeal disease
* Known acute or chronic pancreatitis
* Prior colectomy
* Clinically significant cardiac disease including any of the following:
* CHF requiring treatment (NYHA Classification ≥ 2) in which patients have a history of LVEF < 45% as determined by MUGA scan or ECHO, or uncontrolled hypertension (please refer to WHO-ISH guidelines)
* History or presence of clinically significant ventricular arrhythmias or atrial fibrillation
* Clinically significant resting bradycardia
* Unstable angina pectoris ≤ 3 months prior to starting study drug
* Acute Myocardial Infarction (AMI) ≤ 3 months prior to starting study drug
* QTcF> 480 msec
* Patients with any of the following laboratory values at Screening/baseline:
* Absolute neutrophil count (ANC) <1,500/mm3 [1.5 x 109/L]
* Platelets <100,000/mm3 [100 x 109/L]
* Hemoglobin < 9.0 g/dL
* Serum creatinine>1.5 x ULN
* Serum total bilirubin >1.5 x ULN
* AST/SGOT and/or ALT/SGPT > 2.5 x ULN
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LGX818 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Previous or concurrent malignancy. Exceptions: adequately treated basal cell or squamous cell skin cancer; in situ carcinoma of the cervix, treated curatively and without evidence of recurrence for at least 3 years prior to study entry; or other solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to study entry.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, are not allowed to participate in this study UNLESS they are using highly effective methods of contraception throughout the study and for 3 months after study drug discontinuation. Highly effective contraception methods include:

Total abstinence or

* Male or female sterilization
* Combination of any two of the following (a+b or a+c or b+c)

  1. Use of oral, injected, or implanted hormonal methods of contraception
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

     * Post-menopausal women are allowed to participate in this study. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum Follicle-Stimulating Hormone (FSH) levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Sexually active males must use a condom during intercourse while taking the drug and for 5 T1/2 after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

History of thromboembolic or cerebrovascular events within the last 6 months, including transient ischemic attack, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism.

* Patients who have undergone any major surgery within the last 2 weeks prior to starting study drug or who would not have fully recovered from previous surgery.
* Known Human Immunodeficiency Virus (HIV) infection
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study.
* Treatment with a prior BRAF or MEK inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 07/03/2013 Protocol Closed to Accrual 03/24/2015 Primary Completion Date 03/17/2016 Recruitment Location is the medical clinic
Groups:
- LGX818: Patients With Stage IV or Unresectable Stage III Melanoma Characterized by a BRAFV600 Mutation will receive LGX818 capsules orally on a once -daily schedule (QD) dosing at a dose of 300 mg/day, 2 weeks on followed by a 2 week break. This schedule of 2 weeks on, followed by 2 weeks off, will continue for the duration of time the patients remains on the clinical trial. After the follow up visit patients will be contacted approximately every 12 weeks until they have received a subsequent therapy or until they have been off treatment for a year to monitor their survival.
Period: Overall Study
Arm/Group | LGX818
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LGX818
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 58 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response According to RECIST v1.1 Criteria
Description: Efficacy for all patients will be evaluated by the study sites using RECIST v1.1 and response criteria based on contrast-enhanced CT. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Progression must also involve an increase in size of measurable lesions by at least 5 mm, to minimize the possibility that small changes in a small number of target lesions is falsely interpreted as progression.Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | LGX818
Number analyzed (Participants) | 7
Participants
  Stable Disease | 2
  Partial Response | 2
  Complete Response | 2
  Progressive Disease | 1

2. Secondary Outcome: Response Rate
Description: Response rate (defined as complete + partial response) and 95% confidence interval will be estimated.
Time Frame: 1.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LGX818: LGX818 capsules will be administered orally on a once -daily schedule (QD) dosing at a dose of 300 mg/day, 2 weeks on followed by a 2 week break. This schedule of 2 weeks on, followed by 2 weeks off, will continue for the duration of time the patients remains on the clinical trial. After the follow up visit patients will be contacted approximately every 12 weeks until they have received a subsequent therapy or until they have been off treatment for a year to monitor their survival.
  LGX818
Arm/Group | LGX818
Number analyzed (Participants) | 7
percentage of participants | 57 [20 to 94]

3. Other Pre Specified Outcome: Overall Survival
Description: Overall survival will be calculated for the start of treatment to the date of last death or follow-up.
Time Frame: 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | LGX818
Number analyzed (Participants) | 7
Participants
  Alive | 2
  Dead | 5

4. Other Pre Specified Outcome: Pharmacokinetic (PK) Analysis: Geometric Mean of Maximum Observed Concentration (Cmax) of LGX818 at Steady State
Description: PK parameters will be determined on PK profiles after the first dose and at steady-state using non-compartmental method(s) using WinNonlin
Time Frame: Cycle 1 - Day 1, 15; Cycle 2 - Day 15; Cycle 3 - Day 1, Day 15
Population: Data were not collected
Arm/Group | LGX818
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | LGX818
All-Cause Mortality (participants affected / at risk) | 5/7
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX818 (N=7)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LGX818 (N=7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Arthralgia/myalgia (Musculoskeletal and connective tissue disorders) | 6
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Cutaneous squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bell's Palsy (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
The protocol was stopped after 7 participants were accrued due to intolerable toxicities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes